CLINICAL TRIAL: NCT05418218
Title: International Headache and Vertigo Registration Study
Brief Title: International Headache Registry Study
Acronym: IHRS
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); First People's Hospital of Hangzhou (Other); Affiliated Hospital of Shaoxing Wenli University (Unknown); Tiantai People's Hospital (Unknown); People's Hospital of Lin 'an City (Unknown); Deqing County People's Hospital (Unknown); Jiaxing No.1 Hospital (Unknown); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Shaoxing People's Hospital (Other); Huzhou Central Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Quzhou City People's Hospital (Unknown); Xin Hua Hospital of Zhejiang Province (Other); The First People's Hospital of Huzhou (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); Jiaxing Hospital of Traditional Chinese Medicine (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Linhai First People's Hospital (Unknown); Pain Management Center, Stanford University, USA (Unknown); The Second Affiliated Hospital of Jiaxing University (Other); The Fourth Affiliated Hospital of Medical College of Zhejiang University (Unknown); Chongqing Xinqiao Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20220430
Record Dates: First submitted 2022-04-30; First posted 2022-06-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-10

CONDITIONS: Headache Disorders, Primary; Headache Disorders, Secondary; Migraine; Tension-Type Headache; Vertigo; Vestibular Migraine; Fibromyalgia
Keywords: Migraine; Headache Disorders; Vertigo; Vestibular Migraine; Fibromyalgia
MeSH Terms: conditions — Headache Disorders, Primary; Headache Disorders, Secondary; Migraine Disorders; Tension-Type Headache; Vertigo; Fibromyalgia; Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Migraine: Patients with migraine (including vestibular migraine), including all types of migraine as defined by ICHD-3.
- Other Primary Headache Disorders: Patients with other primary headache disorders (excluding migraine), including all types of other primary headache disorders (such as Tension-Type Headache, Cluster Headache) as defined by ICHD-3.
- Vertigo: Patients with other vertigo disorders (excluding vestibular migraine).
- Secondary Headache Disorders: Patients with secondary headache disorders as defined by ICHD-3.
- Normal control: Normal people do not have headache and vertigo.

SUMMARY:
In the International Headache and Vertigo Registration Study, patients aged 4-99 years with headache (primary headache and secondary headache such as migraine and tension type headache), vertigo (vertigo diseases such as vestibular migraine) and chronic pain (fibromyalgia and other diseases) were collected. The biomarkers, imaging features, right-to-left shunt of the heart (lung), genetic characteristics, treatment, and outcome (in relation to other diseases) of headache-related diseases were studied, and long-term follow-up was planned.

DETAILED DESCRIPTION:
1. Research contents:

   In the International Headache and Vertigo Registration Study, patients aged 4-99 years with headache (primary headache and secondary headache such as migraine and tension type headache), vertigo (vertigo diseases such as vestibular migraine) and chronic pain (fibromyalgia and other diseases) were collected. The biomarkers, imaging features, right-to-left shunt of the heart (lung), genetic characteristics, treatment, and outcome (in relation to other diseases) of headache-related diseases were studied, and long-term follow-up was planned.
2. Research target:

We study biomarkers, imaging features, right-to-left shunt of heart (lung), genetic features, real-world treatment studies, and outcomes (in relation to other diseases) for headache and vertigo related diseases.

ELIGIBILITY:
Inclusion Criteria:

The following are requirements for entry into the study:

1. Written informed consent and participant privacy information (eg, Written Authorization for Use and Release of Health and Research Study Information) obtained from the participant prior to initiation of any study-specific procedures.
2. Male or female participants ages 4 to 99 years, inclusive, at Visit 1.
3. Headache patients meeting the diagnostic criteria for ICHD-3, including primary headaches such as migraine and tension tension-type headaches, secondary headaches, and patients who meet the headache diagnosis in the ICHD-3 appendix (including vestibular migraine).

Exclusion Criteria:

1. Patients who were unable to complete scales such as headache diary.
2. Patients denied or unable to be admitted for long-term follow-up.

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male or female participants ages 4 to 99 years
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2082-12-31 (Estimated); Study Completion 2082-12-31 (Estimated)

PRIMARY OUTCOMES:
Days of Migraine | Medium term: within 6 months after initial diagnosis; long term: 60 years
  The number of days of migraine is the number of days in which migraine occurs or is likely to be migraine (according to IHS ICHD-3 diagnostic criteria).
  A migraine day is a day when a headache lasts for more than 30 minutes, does not take painkillers, and meets the ICHD-3 migraine or most likely migraine criteria. Migraine day can also be defined as a headache day that is effective for the acute treatment of specific migraine drugs (triptan, ditan, gepant, ergotamine, etc.).
Moderate / Severe Headache Days | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Moderate / severe headache days are defined as a day in which moderate or severe pain persists for at least 4 hours, or headache lasts for one day after successful medication for acute headache. These definitions allow the use of relatively simple headache diaries. Subjects were required to indicate whether headache was present (yes / no), peak (mild / moderate / severe) severity and duration (< 4h or 4h), type of acute drug intake (triptan ergot / other), and response to treatment should also be recorded.
Migraine Attack | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Migraine attack is defined as any consistent migraine attacks or the use of specific migraine drugs. If a migraine attack is interrupted by sleep, or temporarily relieved, and then relapses within 48 hours, it is considered an attack. In addition, migraine attacks that were successfully treated with drugs but relapsed within 48 hours and lasted for more than 48 hours were counted as one attack.

SECONDARY OUTCOMES:
The Response Rate of at Least 50%, 75% and 100% Reduction in the Number of Days of Migraine Attacks | Medium term: within 6 months after initial diagnosis; long term: 60 years
  The response rate is calculated as the percentage reduction in the frequency of migraine attacks (or days of migraine, or days of moderate or severe headache) compared with the baseline during each treatment period. The response rate is traditionally defined as a reduction of at least 50% from the baseline, but other percentage reductions (for example: 30%, 75%, 100%) may be used.
Headache Intensity | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Four-point rating scale was used to evaluate the headache intensity of each migraine day--painless, mild, moderate, or severe. Migraine intensity is not recommended as the main outcome measure alone, but it is important to record the decrease in migraine intensity as an indicator of disability reduction.
  Depending on the design of the trial, subjects should be asked to record the intensity of each migraine. In addition, the 11 point visual rating scale (VAS) can be used instead or in combination with the 4-level classification rating scale. The use of VAS in clinical trials may increase the likelihood of showing differences in severity.
Cumulative Hours of Moderate / Severe Pain at 28 Days | Medium term: within 6 months after initial diagnosis; long term: 60 years
  The cumulative number of hours of moderate / severe pain calculated by electronic headache diaries. If an attack occurs before going to bed and when you wake up, the amount of sleep also counts as the number of headache hours.
Days Without Symptoms | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Defined as the number of days without aura, prodromal symptoms, headaches and subsequent symptoms. It needs to be determined by headache diary.
Days Without Headache | Medium term: within 6 months after initial diagnosis; long term: 60 years
  The number of days without headache also includes the number of days without related symptoms directly caused by migraine (including physical function, cognitive or emotional disorders).
Peak Headache Pain Intensity | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Subjects should record the maximum intensity of daily headaches and any medication used. An 11-point digital rating scale can be used instead of or in conjunction with a 4-level classified rating scale.
Migraine Disability Assessment (MIDAS) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  MIDAS is a seven-item questionnaire designed to quantify headache-related disability within 3 months. The MIDAS score is the sum of days of absenteeism or absenteeism caused by headache, days of work or school plus days of housework, days without housework and days without non-work activities caused by headache in the last 3 months.
Headache Impact Scale (HIT-6) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  HIT-6 is a six-question assessment scale used to assess the effects of headache on subjects' ability to work, school, housework and social tasks. The scale assessed the effects of headache on daily life and the functional ability of the subjects. The answer to the evaluation scale is based on the frequency of use of the 5-point scale from "never" to "often". The total score of HIT-6 ranges from 36 to 78, which is the sum of the scores between 6 (never) and 13 (often) for each question.
Migraine Specific Quality of Life Questionnaire (MSQV2.1) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  MSQV2.1 is a 14-item questionnaire used to assess health-related quality of life decline due to migraine in the last 4 weeks. The questionnaire is divided into three areas: the role function limitation area, which is used to assess how migraine restricts the daily social and work-related activities of migraine patients; the role function block area, which is used to assess how migraine prevents these activities; and the emotional function area, which is used to evaluate the emotions associated with migraine. The subjects answered these items using a six-component scale from "never" to "at any time". The original dimension score was calculated by the sum of item answer scores and converted back to 0 to 100. The higher the score, the better the quality of life.
Patient Health Questionnaire (PHQ-9) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  PHQ-9 is a validated, self-administered, concise tool for screening and diagnosis of mental health disorders, which has been tested in office practice. The screening scale is easy to use and can be completed in a short time, which improves the recognition rate of depression and facilitates the diagnosis and treatment of depression. PHQ-9 consists of 9 DSM-Ⅳ diagnostic criteria for depression in the last 2 weeks. Subjects were asked to use a 4-component scale to indicate the frequency of 9 depressive symptoms in the last 2 weeks: 0 (none at all), 1 (a few days), 2 (more than half) and 3 (almost every day). The total score ranges from 0 to 27 (from the best to the worst). A score of 15 to 19 indicates moderate to severe depression and a score of 20 to 27 indicates severe depression.
Generalized Anxiety Disorder (GAD-7) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  GAD-7 is a proven, self-administered and concise tool for screening and diagnosing mental health disorders, which has been tested in the field in office practice. The screening scale is easy to use and can be completed in a short time, which improves the recognition rate of anxiety disorders and facilitates diagnosis and treatment. The main statistical index of this scale is the total score, that is, the sum of item scores. The total score range of GAD-7 is 0: 21 and that of GAD-2 is 0: 6. The score of GAD-7 can be used to evaluate the severity of anxiety symptoms: 0: 4: no clinical significance: anxiety: 5: 9: mild; 10: 14: moderate; > 15: severe. When used as an assistant diagnosis of anxiety symptoms, the cut-off value of GAD-7 is greater than or equal to 10.
Functional Impairment Scale (FIS) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Functional impairment scale (FIS) is a 4-point scale to evaluate the functional status and injury intensity in daily activities. It can be used in conjunction with the four-point pain intensity scale, usually done daily and summarized within four weeks.
Euroqol-5 Dimension Questionnaire (EQ-5D) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  EQ-5D-5Lis a general tool for assessing health status. EQ-5D-5Lconsists of two parts of EQ-5D description system and EQ VAS. The description system consists of five dimensions (activity ability, self-care, daily activities, pain / discomfort and anxiety / depression). Respondents need to tick (or cross) the corresponding boxes of the most appropriate declaration for each of the five dimensions to indicate their health status. The score of the EQ-5D description system generally ranges from 0 (death) to 1 (completely healthy). EQ VAS recorded the respondents' self-rated health outcomes through a vertical visual simulation scale, and the two endpoints were "imaginable ideal health state" and "imaginable least ideal health state". EQ VAS scores range from 0 (the least ideal state of health imaginable) to 100 (the most ideal state of health imaginable).
Suicidal Ideation Score (C-SSRS Scale) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Suicidal ideation should be monitored in trials of central action drugs, higher scores mean a worse outcome.
  Many migraine clinical trials used the Columbia suicide severity scale (C SSRS).The C-SSRS consists of a maximum of 20 items. C-SSRS will be administered in study subjects at each study visit to assess possible suicidal ideation and behavior. Reports of suicidal ideation with intent to act (endorse item 4 or 5) and reports of actual, aborted, or interrupted suicide attempts or a behavior preparatory for making an attempt indicate subjects at high risk for suicide.
Pulse Rate | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Pulse rate will be measured during the visit.It means the number of heartbeats per minute, calculated with a stopwatch.Under normal circumstances, the pulse rate is consistent with the heart rate, and the normal range is 60-100 beats per minute. If it is greater than 100 beats per minute, it is called tachycardia. If it is less than 60 beats per minute, it is called bradycardia.
  Record whether the pulse rate is normal, and describe in detail if abnormal. Record the number of people with clinically significant abnormal pulse rate.
Respiratory Rate | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Respiratory rate will be measured during the visit.It means the number of breaths per minute, calculated with a stopwatch.Clinically, one inhalation and one exhalation are defined as one breath. The normal breathing rate is 12-20 breaths per minute.
  Record whether the respiratory rate is normal, and describe in detail if abnormal.
  Record the number of people with clinically significant abnormal respiratory rate.
Blood Pressure | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Blood Pressure will be measured during the visit，including systolic blood pressure(SBP) and diastolic blood pressure(DBP). It can be calculated with a sphygmomanometer.
  Blood pressure level classification for adults over 18 years old: normal blood pressure (SBP<120 mmHg and DBP<80 mmHg), high normal value [SBP 120-139 mmHg and (or) DBP 80-89 mmHg], hypertension [SBP≥140 mmHg] and (or) DBP≥90 mmHg].
  Record whether the blood pressure is normal, and describe in detail if abnormal.
  Record the number of people with clinically significant abnormal blood pressure.
Body Temperature | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Body temperature will be measured during the visit.It can be calculated with a thermometer.The normal armpit body temperature of an average adult is 36-37°C.
  Record whether the body temperature is normal, and describe in detail if abnormal.
  Record the number of people with clinically significant abnormal body temperature.
Body Mass Index (BMI) | Medium term: within 6 months after initial diagnosis; long term: 60 years
  The following measurements are to be performed: height (initial screening only) and weight. Height and weight are to be measured without shoes. Body Mass Index (BMI) should be calculated using the following formula: BMI (kg/m2= weight (kg)/[height (cm)/100]2.
  A normal BMI is between 20 and 25, over 25 is overweight and over 30 is obese.
Magnetic Resonance Imaging(MRI) T1 | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Patients will accept MRI scans. MRI T1 imaging data and description given by professional radiologist will be collected.
MRI T2 | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Patients will accept MRI scans. MRI T2 imaging data and description given by professional radiologist will be collected.
MRI T2 FLIAR | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Patients will accept MRI scans. MRI T2 FLIAR imaging data and description given by professional radiologist will be collected.
Susceptibility weighted imaging(SWI) in MRI | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Patients will accept MRI scans. SWI imaging data and description given by professional radiologist will be collected.
Arterial spin labeling(ASL) in MRI | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Patients will accept MRI scans. ASL imaging data and description given by professional radiologist will be collected.
Diffusion Tensor Imaging(DTI) in MRI | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Patients will accept MRI scans. DTI imaging data and description given by professional radiologist will be collected.
Echocardiography | Medium term: within 6 months after initial diagnosis; long term: 60 years
  Patients will accept Echocardiography. The degree of Right-to-left Shunt will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Kaiming Liu, Doctor, Principal Investigator — headache specialist clinic of the Second Affiliated Hospital of Zhejiang Medical University
Locations (1):
- Kaiming Liu, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No